CLINICAL TRIAL: NCT07143500
Title: Comparative Study of Action Observation Training Versus Task Oriented Training on Reaching in Patients With Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ahmed Alshimy (Other)
Responsible Party: Sponsor-Investigator, Ahmed Alshimy, Lecturer of Physical Therapy for Neurology and it's Surgery, AlRyada University for Science & Technology
Organization: AlRyada University for Science & Technology (Other)
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: P.T.REC/012/005941
Record Dates: First submitted 2025-08-20; First posted 2025-08-27 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Stroke
Keywords: Stroke; Action Observation Training; Task Oriented Training; Reaching Performance Scale for Stroke; Wolf Motor Function Test
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A (Experimental)
  Interventions: Other: Selected physical therapy program
- Group B (Experimental)
  Interventions: Other: Selected physical therapy program; Other: Task Oriented Training for Upper limb
- Group C (Experimental)
  Interventions: Other: Selected physical therapy program; Other: Action Observation Training Program

INTERVENTIONS:
Other: Selected physical therapy program — Passive stretching, active range of motion exercises, isometric strengthening, and functional gripping practice for the hand
Other: Task Oriented Training for Upper limb — Seated in chair with arm and back support, with forearms resting on a table 73 cm high. Functional movements were trained through task-oriented exercises involving simple activities of daily living(ADL), such as eating (using a plate and spoon), personal hygiene (combing hair, brushing teeth), and tasks using household items (e.g., handling a cup and spoon, or opening a bottle and cap). Each task was repeated five times. Patients were allowed rest periods of five minutes as needed during the exercise sessions.
  Arms: Group B
Other: Action Observation Training Program — sat comfortably in a chair or wheelchair with both arms resting on a table (73 cm high) positioned 50 cm from a 15.6-inch colored laptop screen. They were instructed to attentively observe action videos displayed on the screen and then imitate the observed movements using their affected upper limb. A total of 30 action videos were used, each lasting approximately 50 seconds and demonstrating specific upper limb movements, such as wrist flexion/extension, abduction/adduction, pronation/supination, ulnar/radial deviation, and various grasping and manipulation tasks (e.g., handling coins, pens, a computer mouse, jar lids, bottle caps, typewriting, dialing a phone, and feeding).
  Arms: Group C

SUMMARY:
Stroke is characterized by a sudden onset of localized or generalized brain dysfunction, with symptoms persisting for at least 24 hours or resulting in death. In the chronic phase following a stroke, hand dysfunction is commonly observed, often characterized by reduced finger strength and abnormal hand flexion patterns. Reaching is a crucial aspect of daily tasks, including activities like drinking, interacting with a touch screen, or pressing elevator buttons.

DETAILED DESCRIPTION:
Thirty Nine male chronic stroke patients, aged from 50 to 65 years were included in the study. They were randomly assigned into three equal groups: Group "A" was the control group, Group "B" was the study group I and Group "C" was the study group II). Patients in the control group received a selected physical therapy program for upper limb for 60 minutes, patients in group B received Task Oriented Training for upper limb for 30 minutes and the same selected physical Therapy program for upper limb for 30 minutes, while patients in group C received Action Observation Training for upper limb for 30 minutes and the same selected Physical Therapy Program for upper limb for 30 minutes. The intervention was administered three times weekly over a period of four consecutive weeks. Reaching measurements were done using Reaching Performance Scale for stroke (RPSS) and WolF Motor Function Test (WMFT) pre- and post-treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Chronic stroke diagnosed and referred by a neurologist.
* Patient's ages ranged from 50-65 years old, Duration of stroke was between six to 12 months, Spasticity grade of the upper limb was from 1 to 1+ according to the modified Ashworth scale (MAS).
* Patients with sufficient cognitive abilities that enabled them to understand and follow instructions (Mini-Mental Scale>24), Fugl-Meyer Assessment scale for upper limb scored between 38 and 63.
* Patients with normal vision and hearing, Medically stable patients.

Exclusion Criteria:

* Patients with Upper limb dysfunction due to neurological disorders other than Stroke (e.g, Multiple Sclerosis, Parkinsonism...etc).
* Patients with Severe sensory deficits in the paretic upper limb, Psychological or severe cognitive disorders, Severe cardiovascular disease that can preclude intervention.

Ages: 50 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2025-06-02 (Actual); Primary Completion 2025-07-25 (Actual); Study Completion 2025-08-05 (Actual)

PRIMARY OUTCOMES:
Reaching Performance Scale for Stroke (RPSS) | 4 Weeks
  Evaluates the performance of two reaching and grasping tasks
Wolf Motor Function Test (WMFT) | 4 Weeks
  Designed to assess upper limb motor function following stroke or traumatic brain injury

CONTACTS AND LOCATIONS:
Locations (1):
- Al Ryada University for Science and Technology, Sadat, Menoufia, Egypt

IPD SHARING:
Plan to Share IPD: No